CLINICAL TRIAL: NCT01204489
Title: Lifestyle Intervention for Toddlers at Finnish Welfare Clinics
Brief Title: Lifestyle Intervention for Toddlers Pilot Study
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Tampere University (Other); University of Helsinki (Other); The Finnish Hearth Association (Unknown); The Finnish Food Information (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THL 10109
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensified dietary counseling (Experimental): The dietary intervention consists of tailored dietary counseling, information leaflets and self-evaluation cards given to the families.
  Interventions: Behavioral: Intensified dietary counseling at child wellfare clinics.
- Normal dietary counseling (Active Comparator): Public health nurses continue their usual dietary counseling.
  Interventions: Behavioral: Intensified dietary counseling at child wellfare clinics.

INTERVENTIONS:
Behavioral: Intensified dietary counseling at child wellfare clinics. — The intervention is completed by public health nurses who receive updating education in nutrition. A special training in a family-centred lifestyle counseling method in implemented. The nutrition intervention consists of tailored dietary counseling, information leaflets and self-evaluation card given to the families in the intervention arm. In the control clinics, public health nurses continue their usual dietary counseling.

SUMMARY:
Study aims to pilot a family-centred tailored nutrition intervention at child welfare clinics, targeting the previously observed dietary defaults of Finnish children.

DETAILED DESCRIPTION:
Eating habits can predict diet-related health problems and obesity. The defaults observed previously in the diet of Finnish children include low consumption of vegetables, fruits and vegetable oil-based fats, high consumption of sucrose, poor quality of drinks and low frequency of family meals. Child welfare clinic is the place to promote healthy lifestyles because most Finnish families visit there at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* all families at their child's standard 6-month child welfare clinic visit

Exclusion Criteria:

* families with twins
* families who do not speak Finnish

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To promote child's and family's healthy diet | 8 months
  Changes in family's dietary choices, knowledge and attitudes. Also changes in parent's motivation and self-efficiency to improve family's diet.

CONTACTS AND LOCATIONS:
Overall Officials: Suvi M Virtanen, Professor, Principal Investigator — Head of the Nutrition Unit, professor
Locations (1):
- Child welfare clinics, Espoo, Uusimaa, Finland